CLINICAL TRIAL: NCT06067594
Title: Optimizing Diagnostic Accuracy of Fine Needle Aspiration Biopsy Calcitonin Measurements in Detecting Medullary Thyroid Carcinoma
Brief Title: Calcitonin in Needle Wash Using Electrochemiluminescence Method For Diagnosis Of Medullary Thyroid Carcinoma.
Status: Completed | Type: Observational
Sponsor: Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Maria Julia Cremona, Clinical Professor, Austral University, Argentina
Other Study IDs: 17-042
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Medullary Thyroid Carcinoma; Nodular Goiter
Keywords: calcitonin; calcitonin in washout fluid of fine needle aspiration
MeSH Terms: conditions — Carcinoma, Medullary; Goiter, Nodular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MTC cases: • Cases: Patients who meet the above inclusion and exclusion criteria and have a diagnosis of medullary carcinoma by histology
  Interventions: Diagnostic Test: Fine Needle Aspiration Cytology (FNAC) procedure+calcitonin measurement
- Controls: Controls: Patients who meet the above inclusion and exclusion criteria and do not have a diagnosis of medullary carcinoma by histology.
  Interventions: Diagnostic Test: Fine Needle Aspiration Cytology (FNAC) procedure+calcitonin measurement

INTERVENTIONS:
Diagnostic Test: Fine Needle Aspiration Cytology (FNAC) procedure+calcitonin measurement — Fine needle aspiration (FNA) nodule biopsy: FNA is performed on each patient as long as ATA guideline criteria is met. In case of suspicion of medullary carcinoma, in search of a nodule or medullary focus, FNA will be performed on all non-cystic or spongiform nodules larger than 0.8 cm.
  Other Names: FNA-Ctn

SUMMARY:
Medullary thyroid carcinoma (MTC) is a tumor originating from parafollicular C cells of the thyroid. (1) Representing 1 to 7% of all thyroid carcinoma cases (2, 3, 4). It can occur in two clinical forms, the sporadic or non-hereditary, in 75-80% of patients, and the hereditary form in the remaining 20-25%. It can be part of different clinical syndromes depending on the organs involved: Multiple Endocrine Neoplasia type 2A (MEN2A), Multiple Endocrine Neoplasia type 2B (MEN2B) and Familial Medullary Thyroid Carcinoma (FCM) whose clinical expression is only CMT. A distinctive characteristic of this tumor is its capacity to secrete calcitonin (CT), which, measured in serum, sanctions suspicion of this pathology (5-8) leading to diagnostic studies to confirm CMT. For the preoperative diagnosis of thyroid nodules, ultrasound-guided fine-needle aspiration cytology (FNAC) is a useful and safe procedure; however, its sensitivity to exclude CMT is low (9-15). In 2015, a meta-analysis of 15 studies (16) found that the accuracy of FNAC in diagnosing CMT was around 50%. For this reason, other studies have indicated that the measurement of calcitonin in the fine-needle lavage aspirate fluid of thyroid nodules (CT-guided FNAC), which have suspected medullary carcinoma, can significantly improve the accuracy in the diagnosis of MTC (17 -19). Therefore, clinical practice guidelines recommend its determination in patients with suspected MTC (1,2). The diagnostic importance of pre-surgical medullary carcinoma lies mainly in two points: first, it changes the surgical approach of the patients, and second, it allows one to rule out associated pathologies such as hyperparathyroidism and pheochromocytoma, which are associated when the entity is hereditary. The performance of CT-guided FNAC by the chemiluminescent (CL) method has been widely disseminated. However, to the best of our knowledge, to date there are no data available on the appropriate cut-off value of CT-guided FNAC with calcitonin electrochemiluminescence (ECL) immunometric assay method. As previously stated, it is of particular interest to determine the calcitonin cut-off point in needle washing by electrochemiluminescence method that allows diagnosing medullary carcinoma. Clarifying this point allows improving the approach to patients in whom medullary carcinoma is suspected. This work seeks to determine the cut-off point of CT-guided FNAC for the diagnosis of CMT with the ECL assay method.

DETAILED DESCRIPTION:
Investigative Question:

In daily practice, what value of calcitonin in needle washing by electrochemiluminescent method allows the diagnosis and localization of medullary carcinoma in patients with thyroid nodules with suspected medullary carcinoma? Primary Objective: To determine the cut-off point of calcitonin in fine needle washing of puncture aspiration of thyroid nodules (CT-guided FNA) for diagnosis and localization of medullary carcinoma.Sample Size: Fifty patients with medullary carcinoma and 105 controls will be included. For each case, two controls will be selected, matched by age, sex and non-medullary nodular pathology. In order to estimate the prevalence of medullary carcinoma in patients of the population studied,in whom calcitonin is routinely determined with an accuracy of +/- 2% and a confidence levelof 95%, it is necessary to study 105 patients according to the formula: Study Design: Observational case-control study (patients with medullary carcinoma versus patients without medullary carcinoma). The decision of this design model was due to the low prevalence of medullary carcinoma in the population of patients with thyroid nodules. Methodology: The manuscript followed STARD guidelines for reporting observational and diagnostic studies. Location and Time Period: This multicenter study will be carried out in Argentina including variables obtained from 01.03.2018 to May 31, 2022.Coordinating Institution:- Hospital Universitario Austral: Dr. Cavallo Andrea.- Other study centers invited to participate: Sanatorio Las Lomas San Isidro, and the-Hospital Alta Complejidad Formosa. Dr. Andrea Cavallo will be the principal investigator in the three centers. Patients:A prospective database of patients with punctured thyroid nodules and with serum determination of calcitonin according to the annex presented, as an annex, will be carried out. Patients ≥ 18 years of age, with nodular or multinodular goiter who are undergoing surgery, with normal or elevated serum calcitonin and/or with suspected CMT due to RET mutation from 3/1/2018 to 5/31/2022 will be selected according to inclusion criteria. Patients who do not have a remaining puncture sample, without serum calcitonin, not referred to surgery or those who are lost upon follow-up, will be excluded. The study will be carried out in the Endocrinology Service (Endocrinology area of the Hospital Universitario Austral, Pilar; Hospital Alta Complejidad, Formosa; and Sanatorio Las Lomas, San Isidro). Selection Criteria for Cases and Controls: • Cases: Patients who meet the above inclusion and exclusion criteria and have adiagnosis of medullary carcinoma by histology. • Controls: Patients who meet the above inclusion and exclusion criteria and do not havea diagnosis of medullary carcinoma by histology.For the control group, patients will be randomly selected in a 1:2 ratio, adults, with nodular or multinodular goiter without hypercalcitoninemia, who have surgical criteria. FNA will be performed according to ATA recommendations and with residual sample of FNA washing fluid for calcitonin. It is estimated to include a sample of 100 patients in the control group. Study Variables-Primary Results: The diagnosis of medullary carcinoma is defined according to guidelines of the American Society of Pathologists that uses the Pathological Anatomy service as a diagnostic basis. DATA COLLECTION AND PROCEDURES: In all three institutions the diagnostic work-up of a thyroid nodule includes the combination of personal and family history, physical examination, evaluation of thyroid function, and thyroid US. FNAB is performed following the ATA guidelines recommendations. The data will be obtained from the medical records of the patients (according to authorization requested for the creation of the database) through observation record sheets in Excel (Microsoft). Serum calcitonin test: CT is measured with the same commercially available ECLIA method at the three participating institutions. The determination of calcitonin was carried out on a Cobase601 autoanalyzer with the Elecsys® Calcitonin test (Roche Diagnostics), an electrochemiluminescent immunoassay (ECLIA). As reported by the manufacturer, this test has a detection limit of 0.5 pg/ml, a referenceinterval of up to 9.8 pg/ml for women and 14.3 pg/ml for men, and a measuring range from 0.5to 200,000 pg/ml. Standardization of serum calcitonin sampling and needle washing (in the three institutions) The harmonization of the pre-analytical stage for serum calcitonin determination was ensured in all three centers. This involved morning blood extraction, an 8-hour fasting period, and the collection of fresh serum following laboratory-specific centrifugation protocols. Fresh samples were promptly processed. All centers utilized the same assay for analysis. Evaluation of nodules by ultrasound: All nodules are routinely analyzed in terms of size, echogenicity, number, margin, structure (solid, mixed, or cystic), presence of microcalcifications, and vascularity. According to the ultrasound characteristics, of the American Thyroid Society (ATA). Fine needle aspiration (FNA) nodule biopsy: FNA is performed on each patient as long as ATA guideline criteria is met. In case of suspicion of medullary carcinoma, in search of a nodule or medullary focus, FNA will be performed on all non-cystic or spongiform nodules larger than 0.8 cm. Cytological Analysis: The cytological study will be carried out by expert pathologists, biased to the value of serum Routine Fine Needle Aspiration Cytology (FNAC) procedure: A 23G gauge needle is used under ultrasound guidance. After the smear, the remaining syringe and needle used for washing will be rinsed with 0.5 ml of normal saline. The aspirate will be subjected to calcitonin measurement (all determinations are made in residual fluid sample from the FNA) and will be processed immediately. Definition of hypercalcitoninemia in serum: Female patients with calcitonin levels ≥ 9.8 pg/ml and male patients with calcitonin levels ≥ 14.3 pg/ml. To confirm hypercalcitoninemia, all patients must have at least two serum determinations (it is routinely performed in daily clinical practice as recommended by clinical practice guidelines). The following variables will be verified: a) Inclusion date b) Sexc) Age d) Presentation (nodular or multinodular goiter) e) Number of nodules, location f) Thyroid function (hypothyroidism, hyperthyroidism, Hashimoto's thyroiditis) g) Description of thyroid nodule (echogenicity, margins, consistency, location, presence of calcifications, size) h) Type of thyroid carcinoma (differentiated, medullary, anaplastic, and its variants). Medullary carcinoma was ruled out if Ctn was ≤9.8 pg/mL for women and ≤ 14.3 pg/mL for men, those patients with calcitonin levels ≥ 9,8 pg/mL for women and ≥ 14.3 pg/mL for men and ≤50 pg/mL , were considered as harbouring a low risk for MTC, those with calcitonin ≥ 50 pg/mLl and ≤100 pg/mL, with a moderate risk and those with calcitonin ≥100, with a high risk for MTC 25. In all cases of hypercalcitoninemia, other causes of non-medullary hypercalcitoninemia were ruled-out; first, We repeated serum calcitonin two times throughout the study to minimize the risk of false positives and false negatives attributable to the biochemical test we conducted a comprehensive medical history assessment to identify any underlying conditions that could be responsible for elevated calcitonin levels. This assessment involved using a designed checklist for medications and diseases. To evaluate these conditions, we requested (laboratory tests,. clinical signs, FNA, and pathological examinations).FNAC result (bethesda and cytological description), for each punctured nodule.Pathological anatomy result. TNM and stageSerum calcitonin.Calcitonin in lavage of each punctured nodule. To obtain anatomical, cytological and anatomopathological correlates, each surgical piece was analysed according to the ultrasound data of each patient. Biochemical determinations: TSH, T4l, antithyroid antibodies, calcium, Vit D, PTH, urea, creatinine, clearance, hepatogram, blood count, thyroglobulin.Mortality at last visit Anatomo-pathological analysis: It will be carried out according to standardized norms, in case of doubts or discrepancies they will be resolved internally by three pathologists from each institution. To correlate nodule/spinal focus, an ultrasound correlation (with nodule numbering, cytology, calcitonin in lavage and histology) will be performed in all patients. Possible Biases and Confounding Variables • Selection bias: To avoid this bias in the selection of cases and controls, subjects are followed and treated under the same standards of care. o Cases and controls will be selected by the investigator of the research study (already defined above). • To avoid biochemical determination bias: all determinations will be made using the same procedure, and with the same brand of device. Statistical Analysis Plan For descriptive analysis, continuous variables will be expressed as mean and standard deviation or median and interquartile range (IQR), depending on the observed distribution. The continuous variables were compared by Student's Test for independent samples, one-factor ANOVA or the Mann-Whitney test in case of not complying with the assumptions of normality. To compare qualitative variables, the independence test (Chi-squared) will be used. A clinically relevant cutoff point will be selected to calculate sensitivity, specificity, NPV and PPV and their respective 95% CIs. In all cases, a significance level of less than 5% will be used from the statistical tests applied to reject the hypothesis. The sample will be divided into two groups, those with hypercalcitoninemia, and patients without hypercalcitoninemia that will constitute the control group. ETHICAL ASPECTS The protocol will be sent to the Research Ethics Committee (REC) or Teaching and Research Committee for review and approval. Clinical research will comply with the ethical guidelines indicated in the Declaration of Helsinki of the World Medical Association, in the International Ethical Guidelines for Biomedical Research of the Council for International Organizations of Medical Sciences and in the UNESCO Declaration on Bioethics and Human Rights. (the information cannot be associated, outside of scientific reasons, with a specific person or person. determinable). All data obtained from the study will be handled confidentially and will be available for monitoring if requested by REC participants. If it is necessary to make modifications to what is written in the protocol during the development of the research, new approval will be requested from the REC. The REC can actively monitor the study, ensuring compliance with laws and principles of research ethics. A waiver of informed consent is expected for participating patients beyond that already obtained during medical procedures according to routine practice, since punctures will be performed in nodules larger than 0.8 cm in search of spinal focus in those with hypercalcitoninemia and, in addition, data will be collected from their medical records, according to the request for approval of the creation of the database presented as an annex. This study has no external funding. The selection and inclusion of institutions, data analysis and the results of the different stages of this project will be carried out by the research team described above. Expected Results The determination of the calcitonin cut-off point in needle lavage in patients with thyroid nodules from the general population for the diagnosis of medullary carcinoma is clinically relevant data. Its determination in this population is seldom studied, due to the low incidence of medullary carcinoma in the population of patients with nodular pathology; determining it will allow improvement of the management of patients in daily clinical practice. Therefore, the results are expected to be extremely important for medical science around the world. As mentioned above, there is no work in world literature that determines the cut-off point for calcitonin in lavage in the general population of patients with thyroid nodules for the diagnosis ofm medullary carcinoma. The determination of calcitonin in needle wash is a simple, non-invasive, low-cost method and the results are very precise; and its modulation through the use of a cut-off point has the potential to guide which patients would and would not benefit from a surgical procedure. We believe that this research question will be answered through this multicenter, case control study

ELIGIBILITY:
Inclusion Criteria:Patients ≥ 18 years of age, with nodular or multinodular goiter who are undergoing surgery, with normal or elevated serum calcitonin and/or with suspected CMT due to RET mutation from 3/1/2018 to 5/31/2022 will be selected according to inclusion criteria. -

Exclusion Criteria:Patients who do not have a remaining puncture sample, without serum calcitonin, not referred to surgery or those who are lost upon follow-up, will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a case-control study nested on a prospective multicenter cohort of patients with nodular or multinodular goiter, with normal, or elevated serum Ctn, and thyroidectomy indication.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
medullary carcinoma | 01.03.2018 to May 31, 2022.
  The diagnosis of medullary carcinoma is defined according to guidelines of the American Society of Pathologists that uses the Pathological Anatomy service as a diagnostic basis.
to assess the diagnostic accuracy of FNA-Ctn using an ECLIA for confirmation and localization of MTC, searching for a fixed FNA-Ctn threshold. | 01.03.2018 to May 31, 2022.
  Sensitivity, specificity, and the area under the receiving operator curve (AUROC) were calculated for patients and for the total number of thyroid nodules

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Austral, Pilar, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: data made available ( starting 6 months after publication).
Access Criteria: solicitado por la revista en la cual se publique el artículo

REFERENCES:
- [Result] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Result] Wells SA Jr, Asa SL, Dralle H, Elisei R, Evans DB, Gagel RF, Lee N, Machens A, Moley JF, Pacini F, Raue F, Frank-Raue K, Robinson B, Rosenthal MS, Santoro M, Schlumberger M, Shah M, Waguespack SG; American Thyroid Association Guidelines Task Force on Medullary Thyroid Carcinoma. Revised American Thyroid Association guidelines for the management of medullary thyroid carcinoma. Thyroid. 2015 Jun;25(6):567-610. doi: 10.1089/thy.2014.0335. PMID 25810047
- [Result] Bugalho MJ, Santos JR, Sobrinho L. Preoperative diagnosis of medullary thyroid carcinoma: fine needle aspiration cytology as compared with serum calcitonin measurement. J Surg Oncol. 2005 Jul 1;91(1):56-60. doi: 10.1002/jso.20269. PMID 15999359
- [Result] Kudo T, Miyauchi A, Ito Y, Yabuta T, Inoue H, Higashiyama T, Tomoda C, Hirokawa M, Amino N. Serum calcitonin levels with calcium loading tests before and after total thyroidectomy in patients with thyroid diseases other than medullary thyroid carcinoma. Endocr J. 2011;58(3):217-21. doi: 10.1507/endocrj.k10e-359. Epub 2011 Feb 24. PMID 21358115
- [Result] Boi F, Maurelli I, Pinna G, Atzeni F, Piga M, Lai ML, Mariotti S. Calcitonin measurement in wash-out fluid from fine needle aspiration of neck masses in patients with primary and metastatic medullary thyroid carcinoma. J Clin Endocrinol Metab. 2007 Jun;92(6):2115-8. doi: 10.1210/jc.2007-0326. Epub 2007 Apr 3. PMID 17405835
- [Result] Trimboli P, Mian C, Piccardo A, Treglia G. Diagnostic tests for medullary thyroid carcinoma: an umbrella review. Endocrine. 2023 Aug;81(2):183-193. doi: 10.1007/s12020-023-03326-6. Epub 2023 Mar 6. PMID 36877452
- [Result] Kihara M, Hirokawa M, Kudo T, Hayashi T, Yamamoto M, Masuoka H, Higashiyama T, Fukushima M, Ito Y, Miya A, Miyauchi A. Calcitonin measurement in fine-needle aspirate washout fluid by electrochemiluminescence immunoassay for thyroid tumors. Thyroid Res. 2018 Oct 30;11:15. doi: 10.1186/s13044-018-0059-4. eCollection 2018. PMID 30450128
- [Derived] Cavallo AC, Pitoia F, Roberti J, Brenzoni P, Lencioni M, Jaroslavsky MJ, Spengler E, Voogd A, Firpo C, Saco P, Pinero F, Negueruela M. Optimizing Diagnostic Accuracy of Fine Needle Aspiration Biopsy Calcitonin Measurements in Detecting Medullary Thyroid Carcinoma. Thyroid. 2024 Feb;34(2):186-196. doi: 10.1089/thy.2023.0313. Epub 2024 Jan 12. PMID 38047535